CLINICAL TRIAL: NCT02899546
Title: Suivi Prospectif Des Complications Infectieuses liées Aux PICC Lines en Milieu Tropical
Brief Title: Study of Peripherally Inserted Central Catheter (PICC)-Related Infections in a Tropical Area
Acronym: Septi-PICC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/CHU/Septi-PICC
Record Dates: First submitted 2016-09-07; First posted 2016-09-14 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Catheterization; Peripheral; Infection
Keywords: Peripherally Inserted Central Catheter; Infections; Radiology
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Septi-PICC study aims at assessing incidence of Peripherally Inserted Central Catheter (PICC)-related infections among patients managed in the University Hospital of La Reunion for PICC setting.

DETAILED DESCRIPTION:
Septi-PICC is a prospective single-center study of infections related to PICCs setting at the South tertiary site of the University Hospital of La Reunion over one year with a follow-up of 6 months per patient.

All the complications such as thromboembolic, are collected during the follow-up.

It is planned a convenience sample of 400 patients over 18 years of age, except pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* all patients managed for a PICC setting in the tertiary care hospital

Exclusion Criteria:

* known pregnancy
* minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed for a PICC setting in the tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of PICC-related infections | 1 year with 6 months follow-up

SECONDARY OUTCOMES:
Incidence of other complications following the PICC setting | 6 months follow-up
Incidence of hospitalizations following the PICC setting | 6 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Pierre, France